CLINICAL TRIAL: NCT03459053
Title: CBART: The Reduction of Psychological and Physiological Stress in Women Undergoing IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Soroka University Medical Center (Other); Ben-Gurion University of the Negev (Other); Fondation de Myriam de Senarclens (Unknown)
Responsible Party: Principal Investigator, Johanna Czamanski-Cohen, Lecturer, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CBARTIVF
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Psychological Stress; DNA Degradation, Apoptotic; Telomere Shortening; Fertility Disorders
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research coordinator will conduct the randomization and all information will be deidentified. Investigator will not know who is in which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBART (Experimental): 6 weeks participation in CBART protocol before beginning IVF treatment
  Interventions: Behavioral: CBART
- Wait control (No Intervention): Participants will receive treatment as usual and will be able to receive the intervention after the study is complete.

INTERVENTIONS:
Behavioral: CBART — Cognitive Behavioral protocol that uses art-making for stress reduction and cognitive interventions
  Arms: CBART

SUMMARY:
The study is a randomized controlled trial of a cognitive behavioral interventions and an art-based stress reduction treatment protocol (CB-ART) with 100 women, identified with elevated perceived stress, before undergoing IVF treatment; in order to examine its effect on perceived stress, plasma CFD, telomere length and pregnancy rates.

CB-ART is a 6-session treatment protocol that has been utilized with women coping with stress, depression and pain and is effective in reducing these indicators, developed and evaluated by our research team. The treatment protocol emphasizes processing together with the client's recalled image, symptom or memory (ISM) pertaining to a current distressing mental or physical state. CB-ART is a multi-method model that integrates cognitive behavioral interventions and art-based stress reduction interventions. The innovation in this method is the transformation of imagined and drawn images and memories rather than solely verbally discussing their contents. The focus is on changing compositional elements that comprise each image and memory, thus providing a therapeutic venue to reframe and transform stress producing, recalled images and memories and reduce symptoms of perceived stress. Art making is beneficial for eliciting an emotional response and provides a concrete platform to conduct the cognitive processing that initiate change on the paper and then in the mind. Furthermore, the soothing qualities of interacting with art making foster and enhance behavioral relaxation techniques.

Our study population, women with infertility problems, who are designated to undergo IVF treatment and have been identified to have elevated perceived stress scores on the Perceived Stress Scale (above 15) will be randomized and allocated to receive the CB-ART intervention tailored to reduce stress or treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking nulliparous women
* between the ages of 18-35
* without an axis I psychiatric diagnosis

Exclusion Criteria:

* Women over 35
* Do not speak Hebrew
* Have an Axis I psychiatric diagnosis that would prevent them from participating in the intervention

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | 2 months
  The perceived stress scale (Cohen, Kamarck & Mermelstein, 1994) is a 10 item scale measuring perceived stress by asking 10 questions in which participants are requested to list on a scale from 0- never to 4- very frequently, how often they have experienced different stress related occurrences in the past month. The scale is calculated by summing the items (4 items reversed) with scores ranging from 0 - 40. Higher scores indicate higher perceived stress, with the mean US score being 16.

SECONDARY OUTCOMES:
Cell Free DNA | 2 months
  DNA particles outside the cell nuclous as found in plasma
Telomerase | 2 months
  Enzyme related to telomere length, as found in PMBC
Pregnancy | 2 months
  hCG levels higher than 8 in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Harvardi, PhD, Principal Investigator — Soroka University Medical Center; Julie Cwikel, PhD, Principal Investigator — Ben-Gurion University of the Negev; Orly Sarid, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czamanski-Cohen J, Sarid O, Cwikel J, Levitas E, Lunenfeld E, Douvdevani A, Har-Vardi I. Decrease in cell free DNA levels following participation in stress reduction techniques among women undergoing infertility treatment. Arch Womens Ment Health. 2014 Jun;17(3):251-3. doi: 10.1007/s00737-013-0407-2. Epub 2014 Jan 14. PMID 24420416
- [Background] Czamanski-Cohen J, Sarid O, Cwikel J, Lunenfeld E, Douvdevani A, Levitas E, Har-Vardi I. Increased plasma cell-free DNA is associated with low pregnancy rates among women undergoing IVF-embryo transfer. Reprod Biomed Online. 2013 Jan;26(1):36-41. doi: 10.1016/j.rbmo.2012.09.018. Epub 2012 Oct 4. PMID 23182744
- [Background] Czamanski-Cohen J, Sarid O, Cwikel J, Douvdevani A, Levitas E, Lunenfeld E, Har-Vardi I. Cell-free DNA and telomere length among women undergoing in vitro fertilization treatment. J Assist Reprod Genet. 2015 Nov;32(11):1697-703. doi: 10.1007/s10815-015-0581-4. Epub 2015 Oct 5. PMID 26438644
- [Background] Sarid O, Cwikel J, Czamanski-Cohen J, Huss E. Treating women with perinatal mood and anxiety disorders (PMADs) with a hybrid cognitive behavioural and art therapy treatment (CB-ART). Arch Womens Ment Health. 2017 Feb;20(1):229-231. doi: 10.1007/s00737-016-0668-7. Epub 2016 Sep 19. PMID 27645306